CLINICAL TRIAL: NCT03536923
Title: Use of the Leva Incontinence System in Treating Bladder Incontinence.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Renovia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REN-01
Record Dates: First submitted 2018-05-13; First posted 2018-05-25 (Actual); Results first posted 2018-12-12 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Stress Urinary Incontinence
Keywords: Female
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Leva Arm (Experimental): Subjects will use the leva device twice daily to perform pelvic floor muscle exercises
  Interventions: Device: Leva Incontinence System For Pelvic Floor Muscle strengthening

INTERVENTIONS:
Device: Leva Incontinence System For Pelvic Floor Muscle strengthening — The leva device is placed vaginally for 2.5 minutes twice daily, and pelvic floor muscle exercises are performed based on guidance from data sent from the device to their mobile phone.

SUMMARY:
This open-label proof-of-concept study is designed to evaluate the impact of the leva digital incontinence system on the treatment of stress and mixed urinary incontinence in women over a six week period. Subjects will participate in a 2.5 minute exercise program twice daily (performed at a clinic with therapist assistance 5x weekly, and at home once daily on weekdays and twice daily on weekends. Validated surveys (UDI-6, IIQ-7 and PGI-I) will be used to evaluate symptom relief. A battery of pelvic floor muscle exercises will be performed weekly to evaluate progress in muscle strengthening.

ELIGIBILITY:
Inclusion Criteria

* Subjects must be female.
* Subjects must be capable of giving informed consent.
* Subjects should be at least 18 years of age and less than 89 years of age
* Subjects must have a diagnosis of or symptoms of predominant mild to moderate urinary incontinence based on the results of the completed urinary incontinence surveys.

Exclusion Criteria:

* Absence of a vagina.
* Positive drug or alcohol test at the screening visit.
* Post-menopausal defined as absence of a period for over 12 months.
* Pregnancy or being less than 12 months post-partum.
* Greater than three vaginal deliveries or prior operative delivery (e.g. use of vacuum, forceps or abdominal pressure).
* Symptoms of stage II or greater pelvic organ prolapse.
* BMI >31 kg/m2.
* Diagnosis of any neurological disorder.
* Prior lower back or pelvic surgery, including prior surgery for stress urinary incontinence (SUI).
* Prior pelvic radiation.
* Current or recurrent vaginal infections (>three per year).
* Painful bladder syndrome, active or chronic pelvic pain.
* Concurrent Pelvic Floor Muscle Exercises (PFME) under a supervised therapeutic plan of care.
* Previous supervised pelvic floor muscles rehabilitation in the past 12 months for the treatment for urinary incontinence or any other pelvic floor disorder.
* Currently taking medication to treat incontinence.
* Impaired cognitive function.
* Unable to tolerate use of the leva device.

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Subject must have a vagina
Enrollment: 23 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2017-08-12 (Actual); Study Completion 2017-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Rosenberg, MD, Principal Investigator — New England Spine Center
Locations (1):
- New England Spine Center, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Leva Arm
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Leva Arm: Subjects will use the leva device twice daily to perform pelvic floor muscle exercises
  Leva Incontinence System For Pelvic Floor Muscle strengthening: The leva device is placed vaginally for 2.5 minutes twice daily, and pelvic floor muscle exercises are performed based on guidance from data sent from the device to their mobile phone. Subjects completed one daily exercise under direct supervision 5x weekly. The remaining daily exercise on weekdays, and twice daily on weekends, were performed at home at the subject's discretion.
Arm/Group | Leva Arm
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 17
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 23
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26 (4)
Parity [Count of Participants; unit: Participants]
  Births=0 | 6
  Births=1 | 5
  Births=2 | 10
  Births=3 | 2

OUTCOME MEASURES:

1. Primary Outcome: Symptoms of Urinary Incontinence at Baseline and at 6 Weeks
Description: A validated, standardized questionnaire (the short form of the urogenital distress inventory, UDI-6) will be used to evaluate change in symptoms of urinary incontinence. Minimum score = 0, Maximum score = 100, lower scores indicate fewer symptoms.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Leva Arm
Number analyzed (Participants) | 23
score on a scale
  Baseline | 27.5 (16.9)
  Final (week 6) | 1.1 (2.9)
Statistical Analysis 1: Comparison: Leva Arm; Test type: Other; p = 0.0001, t-test, 1 sided

2. Secondary Outcome: Condition-specific Quality of Life Assessment (IIQ-7) at Baseline and 6 Weeks.
Description: Condition specific quality of life as it is affected by urinary incontinence will be assessed using the Incontinence Impact Questionnaire (IIQ-7). Minimum value 0, Maximum value 100, lower scores indicate improvement.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Leva Arm
Number analyzed (Participants) | 23
score on a scale
  Baseline | 17.6 (21.6)
  Final (week 6) | 0.2 (1.0)
Statistical Analysis 1: Comparison: Leva Arm; Test type: Other; p = 0.0009, t-test, 1 sided

3. Secondary Outcome: Number of Participants for Different Categories of Patient Global Impression of Improvement (PGI-I)
Description: Subject perception of improvement will be evaluated using the standardized survey Patient Global Impression of Improvement (PGI-I). Categories of improvement include: Very Much Better, Much Better, A Little Better, No Change, Worse(any degree).
Time Frame: At 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Leva Arm
Number analyzed (Participants) | 23
Participants
  Very Much Better | 17
  Much Better | 4
  A Little Better | 2
  No Change | 0
  Worse, Any Degree | 0

4. Secondary Outcome: Pelvic Floor Muscle Performance (Mean Maximum Duration of Voluntary Pelvic Floor Muscle Contraction)
Description: Change in pelvic floor muscle performance will be evaluated using muscle performance testing performed using the leva device. Subjects were asked to lift and squeeze pelvic floor muscles for as long as possible. The length of time a subject can "hold" the lift was recorded
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Leva Arm
Number analyzed (Participants) | 23
seconds
  Baseline | 13 (12)
  Final (week 6) | 187 (46)
Statistical Analysis 1: Comparison: Leva Arm; Test type: Other; p = 0.0001, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a 6-week period
Arm/Group | Leva Arm
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 3/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leva Arm (N=23)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Common Cold
Suspected urinary tract infection (Renal and urinary disorders) | 1 (1) — Culture negative irritative voiding
Migraine Headache (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This is a single-arm, proof of concept trial. As such it lacks a comparison arm, planned in future studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-14): https://cdn.clinicaltrials.gov/large-docs/23/NCT03536923/Prot_SAP_000.pdf